CLINICAL TRIAL: NCT05400070
Title: A Single-arm Clinical Study to Investigate the Efficacy and Safety of Neoadjuvant PD-1 Inhibitor (Sintilimab), Anlotinib Combined With Chemotherapy in Resectable Stage IIA-IIIB NSCLC
Brief Title: Neoadjuvant PD-1 Inhibitor (Sintilimab), Anlotinib Combined With Chemotherapy in Resectable Stage IIA-IIIB NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K202104-03
Record Dates: First submitted 2022-05-18; First posted 2022-06-01 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Sintilimab; Lung Cancer; Anlotinib; Chemotherapy
Keywords: Sintilimab, Anlotinib. chemotherapy. safety. efficacy
MeSH Terms: conditions — Lung Neoplasms | interventions — anlotinib; Drug Therapy; sintilimab

STUDY DESIGN:
Intervention Model Description: Sintilimab (200mg fixed dose) iv, d1, q3w + anlotinib 10mg, po, qd1-14, q3w, was evaluated after 3 cycles of chemotherapy and stopped for 3 weeks (21 days) after surgery for 4-6 weeks (21-42 days) after the last dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- neoadjuvant therapy (Experimental): Sintilimab (200mg fixed dose) iv, d1, q3w，anlotinib 10mg, po, qd1-14, q3w combine with Chemotherapy
  Interventions: Drug: Neoadjuvant therapy 1

INTERVENTIONS:
Drug: Neoadjuvant therapy 1 — Dosing regimen Sintilimab (200mg fixed dose) iv, d1, q3w + anlotinib 10mg, po, qd1-14, q3w, was evaluated after 3 cycles of chemotherapy and stopped for 3 weeks (21 days) after surgery for 4-6 weeks (21-42 days) after the last dose.
  Other Names: anlotinib 10mg, po, qd1-14, q3w; Chemotherapy; Sintilimab (200mg fixed dose) iv, d1, q3w

SUMMARY:
primary purpose：Observe the pathological complete response rate (PCR) of postoperative tumor tissue resection and evaluate the safety of the treatment process.

DETAILED DESCRIPTION:
primary purpose：Observe the pathological complete response rate (PCR) of postoperative tumor tissue resection and evaluate the safety of the treatment process.

Description of the study design This is a single-center, prospective, open-label, single-arm clinical study to preliminarily explore the single-arm clinical study administration and drug management of Sintilimab, anlotinib combined with neoadjuvant chemotherapy in stage IIA-IIIB NSCLC

Dosing regimen Sintilimab (200mg fixed dose) iv, d1, q3w + anlotinib 10mg, po, qd1-14, q3w, was evaluated after 3 cycles of chemotherapy and stopped for 3 weeks (21 days) after surgery for 4-6 weeks (21-42 days) after the last dose.

ELIGIBILITY:
Inclusion Criteria:

1. pathological diagnosis of lung cancer, Age 18 years and 75 years old, physical strength status score 0-1;
2. The investigator believes that the subject can comply with the study protocol;
3. The investigator has confirmed to have at least one measurable lesion according to the RECIST1.1 criteria;
4. Stage IIA, IIB, IIIA, IIIB NSCLC with histological or cytology proven operable treatment according to the International Association for Lung Cancer Research and the American Joint Committee on Cancer Staging version 8;
5. Good hematopoietic function, defined as absolute neutrophil number 1.5X109 / L (no granulocyte colony stimulating factor support therapy), platelet count 100X109 / L, hemoglobin 90 g / L; (no transfusion or no erythropoietin dependence within 7 days);
6. Good liver function, defined as 1.5 times the normal limit (ULN) of serum total bilirubin; ULN at 2.5 times transaminase (AST) and ALT); AST and ALT for recorded ULN;
7. Good renal function, defined as serum creatinine 1.5 times ULN or calculated creatinine clearance of 60 ml/min (Cockcroft-Gault formula); routine urine protein less than 2 +, or 24h urine protein <1g;
8. Good coagulation function, defined as the international standardized ratio (INR) or prothrombin time (PT) 1.5 times ULN;
9. The total amount of lung function (e. g., FVC, FEV1, TLC, FRC, and DLco) can tolerate the proposed lung resection procedure;
10. For female subjects of childbearing age, the urine or serum pregnancy test should be negative within 3 days before receiving the first dose (cycle 1, day 1)

Exclusion Criteria:

1 . Presof locally advanced unresectable or metastatic disease;

2.. peripheral neuropathy;

3.Active, known or suspected autoimmune diseases, type I diabetes, hypothyroidism that requires only hormone replacement therapy, skin diseases that do not require systemic treatment (such as vitiligo, psoriasis or alopecia), or diseases not expected to recur without external stimulus factors can be selected;

4. Systemic treatment with corticosteroids (an equivalent dose of> 10 mg prednisone per day) or other immunosuppressive drugs within 14 days before randomization.Inhalor topical steroids are permitted without active autoimmune disease.

5.Active Hepatitis B / hepatitis C infection and known HIV;

6.Patients who have previously received chemotherapy or any other anti-tumor therapy;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (PCR) | up to 4 months
  pathological complete response (PCR)

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, the Air Force Military University, Xi'an, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Duan H, Shao C, Luo Z, Wang T, Tong L, Liu H, Yao X, Lei J, Zhao J, Gao Y, Jiang T, Yan X. Perioperative sintilimab and neoadjuvant anlotinib plus chemotherapy for resectable non-small-cell lung cancer: a multicentre, open-label, single-arm, phase 2 trial (TD-NeoFOUR trial). Signal Transduct Target Ther. 2024 Oct 28;9(1):296. doi: 10.1038/s41392-024-01992-0. PMID 39465257